CLINICAL TRIAL: NCT06737796
Title: The Effect of Different Feeding Methods on Infant's Weight, Full Oral Feeding Transition Time and Success of Breastfeeding in Preterm Infants
Brief Title: The Effect of Different Feeding Methods on Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Tugba Yapar, Principal investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Adnan Menderes Univercity
Record Dates: First submitted 2024-01-17; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Preterm Infants; Injector; Finger; Sucking Success; Nursing Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental 1 (Experimental): Preterm babies in the finger feeding group, which constituted the study group, were finger fed by the neonatal intensive care nurse responsible for the baby's care, three times a day for no more than 20 minutes. If babies had breast milk during feedings, breast milk was given first. Formula milk was used when breast milk was not available. The amount of milk that the preterm baby should receive, determined by the neonatal specialist physician, was completed after the planned 20 minutes of feeding time and at other feeding meals during the day, according to the clinic's feeding protocol. In addition, preterm babies have three meals a day; Heart rate, respiration and saturation before and after feeding, and evaluation of feeding duration, amount of feeding and vomiting at the end of feeding were recorded in PBIF. The Preterm Baby Monitoring Form, which was planned to be used at this stage, was filled out by the neonatal intensive care nurse or the researcher.
  Interventions: Behavioral: Finger Feeding
- experimental 2 (Experimental): Preterm babies in the syringe feeding group, which constituted the other study group, were fed with a syringe three times a day for no more than 20 minutes by the neonatal intensive care nurse responsible for the baby's care. If babies had breast milk during feedings, breast milk was given first. Formula milk was used when breast milk was not available. The amount of milk that the preterm baby should receive, determined by the neonatal specialist physician, was completed after the planned 20 minutes of feeding time and at other feeding meals during the day, according to the clinic's feeding protocol. In addition, preterm babies have three meals a day; Heart rate, respiration and saturation before and after feeding, and evaluation of feeding duration, amount of feeding and vomiting at the end of feeding were recorded in PBIF. The Preterm Baby Monitoring Form, which was planned to be used at this stage, was filled out by the neonatal intensive care nurse or the researcher.
  Interventions: Behavioral: syringe feeding

INTERVENTIONS:
Behavioral: Finger Feeding — feeding method
  Arms: experimental 1
Behavioral: syringe feeding — feeding method
  Arms: experimental 2

SUMMARY:
Objective: The aim of this study was to investigate the effect of finger feeding and syringe feeding methods on infant weight, time to full oral feeding and breastfeeding success in preterm infants.

H01: There is no difference between the weights of preterm babies fed by finger and by syringe.

H02: There is no difference in the transition time between finger-fed and syringe-fed preterm babies to full oral feeding.

H03: There is no difference between breastfeeding success between finger and syringe feeding methods.

DETAILED DESCRIPTION:
The study was conducted as a parallel groups randomized experimental study. The study was conducted between December 1, 2021 and June 1, 2023 in the Neonatal Intensive Care Unit of Aydın Obstetrics and Gynecology Hospital. The sample included preterm infants with 320/7-366/7 gestation weeks who were receiving care and treatment in the neonatal intensive care unit. In the sample, n=38 infants were randomly assigned to study group 1 and n=36 infants to study group 2 and the study was completed with n=74 infants. The data were collected using the Preterm Infant Information Form, Preterm Infant Follow-up Form and LATCH Breastfeeding Diagnostic Measurement Tool. The babies selected for the study group were fed with the method of whichever study group they were added to (finger or syringe feeding) at three feeding meals each day. After switching to full oral feeding, breastfeeding success was measured with the breastfeeding diagnostic measurement tool (LATCH), which was used when the infants first held the breast and the time of transition to full oral feeding. The difference between groups was analyzed using Mann Whitney U analysis for non-normally distributed data and the difference between groups for normally distributed data was analyzed using independent two sample t test. Homogeneity of variances was assessed by Levene's test. Since the standard error indicates the spread of the means of the samples selected from the same population and the standard deviation indicates the distance of each individual in the group from the mean, the standard error values were given together with the means in the analyses comparing the group means.

ELIGIBILITY:
Inclusion Criteria:

* Having a gestational age between 32 weeks and 36+6 weeks,
* Weighing 1500 g or more,
* Having spontaneous breathing (can receive free oxygen, incubator oxygen),
* Those who have been fed only by gavage or parenterally and are ready to switch to oral feeding,
* Preterm babies whose parents were literate in Turkish and gave consent were included in the study.

Exclusion Criteria:

* Those who were fed orally before the research,
* Those who need noninvasive mechanical ventilation such as CPAP,
* Babies with metabolic diseases were excluded from the study.

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Mother and Preterm Baby Introductory Information Form (APBTBF): | avarege four days
  Mother and Preterm Baby Introductory Information Form (APBTBF): The questionnaire prepared by the researcher in line with the literature includes introductory information about the preterm baby (delivery type, baby's birth date and time, hospitalization date and time, hospitalization diagnosis, gestational age, corrected gestational age, gender). , birth weight, birth length, birth head circumference, weight at the start of the study, birth order, whether the mother was breastfed or not, whether the mother was educated about expressing her milk, discharge weight, date and time of the baby's discharge from the hospital) and descriptive information about the mother (age, education). It consists of 22 questions asking about breastfeeding level, previous breastfeeding experience, breastfeeding duration if breastfeeding, and previous birth to a preterm baby).
Preterm Baby Follow-up Form (PBIF): | avarege four days
  Preterm Baby Follow-up Form (PBIF): It is a follow-up form developed by the researcher in line with the literature in order to follow the preterm baby from the moment he starts feeding with an alternative feeding method. In this form, the preterm baby's birth, transition to oral feeding, transition to breastfeeding and discharge dates, as well as information on body weight, head circumference and height at these stages; Information on heart rate (HR), respiratory rate and oxygen saturation (SpO2) values before and after feeding, presence of vomiting after feeding, full oral feeding amounts and feeding durations are included.
Breastfeeding Diagnostic Measurement Tool (LATCH): | avarege four days
  Breastfeeding Diagnostic Measurement Tool (LATCH): LATCH was developed by Deborah Jensen and Sheilla Wallace in 1993. The adaptation of the scale into Turkish and its validity and reliability studies were first carried out in a Master's Thesis study by Demirhan and Pek in 1997, but this study was not published. The second validity and reliability study was conducted by Yenal and Okumuş in 2003. In the application of the scale, the mother is observed by a midwife/nurse while breastfeeding, and the form is filled out by evaluating the mother and the baby in line with the criteria. The application time of the scale is 5-10 minutes. While the Cronbah alpha value of the original version of the vehicle was found to be 0.93, it was found to be 0.95 in the Turkish adaptation study. The measurement tool consists of five evaluation items/criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes Univercity, Aydin, efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No